CLINICAL TRIAL: NCT06226207
Title: Validity and Reliability of Turkish Version of Physiotherapy Mobile Acceptance Questionnaire
Brief Title: Mobile Acceptance Questionnaire in Physiotherapy
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, Karabuk University
Other Study IDs: Questionnaire
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Reliability and Validity
Keywords: Mobile Health Apps; Physiotherapy Mobile Acceptance Questionnaire; Health; Technology assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many studies were conducted on the determinants and acceptance of mobile or wearable health care technology (mHealth). However, little research was done on physiotherapists' thinking regarding the use of mHealth. In this study, it was aimed to test the suitability of the Physiotherapy Mobile Acceptance Questionnaire -PTMAQ which was developed by Blumenthal et al. [6] to evaluate the physiotherapists' Perspectives on the Use of Mobile or Wearable Technology in their clinical practice, to the assessments of physiotherapists (to understand attitudes and possible barriers). PTMAQ, based on the Technology Acceptance Model (TAM) by Blumenthal et al. [6] was translated into Turkish and applied to Physiotherapists working in Turkey. Thus, it is expected that the results to be obtained after the scale is applied in Turkish language and in the Turkish sample will contribute to the further development of the scale. In this respect, the study is important both in terms of bringing a new PTMAQ to the literature and making suggestions to researchers and academicians who will use this scale in the future.

DETAILED DESCRIPTION:
Due to the necessity of collecting data from a large sample to test the research's hypotheses, the questionnaire was chosen as the data collection instrument. The Physiotherapy Mobile Acceptance Questionnaire (PTMAQ) scale developed by Blumenthal et al. [6] was translated into Turkish and used for data collection on the variables of the study. In this scale, it was seen that a total of 8 expressions belonging to the Perceived usefulness (4 expressions) and Perceived ease of use (4 expressions) variables were used by making use of the TAM model to reveal the attitudes of the participants (physiotherapist) that could affect their intentions towards mHealth practice. Then, a question consisting of 4 statements was asked to reveal the effect of these variables on the intention to use of early adopters. Finally, 18 statements were used to measure the effect of intention to use on intention/likelihood to recommend an mHealth tool for specific clinical purposes.

Based on the clinical usefulness of MWT, these 18 statements want to determine the probability of physiotherapists recommending MWT to patients based on the clinical usefulness of using MWT in 3 dimensions (gait speed, gait quality and balance, pain/cognitive status). Responses were requested in a 5-point Likert format to the statements in the scale, according to which "1=Strongly Disagree" means "5=Strongly Agree". For the scale adaptation procedure, Blumenthal et al., the creators of the PTMAQ scale, were contacted via email and permission was secured. After that, five academics who had an excellent command on English translated it into Turkish. Attempts were made to establish language validity using the back translation technique. It was translated into the target language by an expert in the field of English, and the similarity was determined by translating it from the target language into English. Consequently, it was determined that the forms created independently in the two languages are comparable. Before conducting field research, a draft questionnaire was administered to forty physiotherapists, who were then interviewed face-to-face about concepts and expressions. In this manner, the potential miscommunication-causing wording errors in the questionnaire were reviewed, and the questionnaire was finalized.

ELIGIBILITY:
Inclusion Criteria:

* Having completed at least 4 years of physiotherapy and rehabilitation education at undergraduate level and having the title of physiotherapist.
* Being actively practicing their profession in universities, hospitals, rehabilitation centers, etc.
* Being able to communicate in Turkish
* Volunteering to participate in the study

Exclusion Criteria:

-

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 421 physiotherapists will be included in the research.
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Physiotherapy Mobile Acceptance Questionnaire (PMAQ) | First Day
  It is a survey consisting of 30 questions examining physiotherapists' adoption behaviors on mobile health. It consists of 12 items assessing adoption of technological applications and 18 items related to clinical variables for which mHealth technology can be recommended. Clinical variables in this context consist of (1) general activity level, (2) balance, (3) walking speed, (4) walking quality, (5) cognitive status and (6) pain. There are 5 answer options for each question, including: strongly disagree, disagree, undecided, agree, and strongly agree (6).
  Additionally, following the survey, individuals' demographic information and smartphone ownership and usage status will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Metehan YANA PhD, Principal Investigator — Karabuk University
Locations (1):
- Karabük University, Karabük, Turkey (Türkiye)

REFERENCES:
- [Background] Gagnon MP, Orruno E, Asua J, Abdeljelil AB, Emparanza J. Using a modified technology acceptance model to evaluate healthcare professionals' adoption of a new telemonitoring system. Telemed J E Health. 2012 Jan-Feb;18(1):54-9. doi: 10.1089/tmj.2011.0066. Epub 2011 Nov 14. PMID 22082108
- [Background] Palos-Sanchez PR, Saura JR, Rios Martin MA, Aguayo-Camacho M. Toward a Better Understanding of the Intention to Use mHealth Apps: Exploratory Study. JMIR Mhealth Uhealth. 2021 Sep 9;9(9):e27021. doi: 10.2196/27021. PMID 34499044
- [Background] Hoque R, Sorwar G. Understanding factors influencing the adoption of mHealth by the elderly: An extension of the UTAUT model. Int J Med Inform. 2017 May;101:75-84. doi: 10.1016/j.ijmedinf.2017.02.002. Epub 2017 Feb 10. PMID 28347450
- [Background] Blumenthal J, Wilkinson A, Chignell M. Physiotherapists' and Physiotherapy Students' Perspectives on the Use of Mobile or Wearable Technology in Their Practice. Physiother Can. 2018 Summer;70(3):251-261. doi: 10.3138/ptc.2016-100.e. PMID 30275650
- [Background] Rai A, Chen L, Pye J, Baird A. Understanding determinants of consumer mobile health usage intentions, assimilation, and channel preferences. J Med Internet Res. 2013 Aug 2;15(8):e149. doi: 10.2196/jmir.2635. PMID 23912839